CLINICAL TRIAL: NCT05346484
Title: A Phase I, Dose Escalation Safety and Tolerability Study of VAXINIA (CF33-hNIS), Administered Intratumorally or Intravenously as a Monotherapy or in Combination With Pembrolizumab in Adult Patients With Metastatic or Advanced Solid Tumors (MAST).
Brief Title: A Study of CF33-hNIS (VAXINIA), an Oncolytic Virus, as Monotherapy or in Combination With Pembrolizumab in Adults With Metastatic or Advanced Solid Tumors
Acronym: MAST
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CF33-hNIS-002
Record Dates: First submitted 2022-03-22; First posted 2022-04-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Solid Carcinoma; Solid Tumor, Adult; Metastatic Cancer; Advanced Solid Tumor; Cholangiocarcinoma; Bile Duct Cancer
Keywords: oncolytic virus
MeSH Terms: conditions — Neoplasm Metastasis; Cholangiocarcinoma; Bile Duct Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CF33-hNIS IT Administration Monotherapy (Experimental)
  Interventions: Biological: CF33-hNIS
- CF33-hNIS IV Administration Monotherapy (Experimental)
  Interventions: Biological: CF33-hNIS
- CF33-hNIS IT Administration in Combination with Pembrolizumab (Experimental)
  Interventions: Biological: CF33-hNIS; Biological: Pembrolizumab
- CF33-hNIS IV Administration in Combination with Pembrolizumab (Experimental)
  Interventions: Biological: CF33-hNIS; Biological: Pembrolizumab
- CF33-hNIS IV Administration in Combination with modified FOLFOX (Experimental)
  Interventions: Biological: CF33-hNIS; Drug: Modified FOLFOX

INTERVENTIONS:
Biological: CF33-hNIS — CF33-hNIS is a chimeric orthopoxvirus (oncolytic virus) engineered to express the human sodium iodide symporter (hNIS)
  Other Names: VAXINIA; HOV2
Biological: Pembrolizumab — Pembrolizumab 200mg administrated IV every 3 weeks (Q3W).
  Other Names: KEYTRUDA®
  Arms: CF33-hNIS IT Administration in Combination with Pembrolizumab; CF33-hNIS IV Administration in Combination with Pembrolizumab
Drug: Modified FOLFOX — 28 day cycle of:
  * Leucovorin calcium/folinic acid
  * Fluorouracil
  * oxaliplatin
  Arms: CF33-hNIS IV Administration in Combination with modified FOLFOX

SUMMARY:
This is an open-label, dose-escalation, multi-center phase I study evaluating the safety of CF33-hNIS (hNIS - human sodium iodide symporter) administered via two routes of administration, intratumoral (IT) or intravenous (IV), either as a monotherapy or in combination with pembrolizumab or mFOLFOX in patients with metastatic or advanced solid tumors.

DETAILED DESCRIPTION:
CF33-hNIS, a novel chimeric orthopoxvirus, will be administered as a monotherapy or in combination with pembrolizumab or mFOLFOX to assess the safety and efficacy of the treatment regimens as well as immunological changes in the tumour microenvironment.

Patients eligible for treatment in dose escalation IT/IV cohorts include those with any metastatic or advanced solid tumor who have documented radiological progression per RECIST following at least two prior lines of therapy which may have included treatment with an Immune Checkpoint Inhibitor(ICI). For expansion IT and IV cholangiocarcinoma cohort patients, one prior line of systemic chemotherapy in metastatic/advanced setting is required and for patients with targetable tumor mutations, must have also received 1 line of an approved targeted therapy. For expansion IV cholangiocarcinoma cohort, prior treatment with leucovorin calcium, fluorouracil, or oxaliplatin is not permitted.

For IT/IV cohorts, patients will be treated with CF33-hNIS on Day 1 and 8 of Cycle 1 and then on Day 1 of each cycle thereafter. Patients treated with the combination regimen with pembrolizumab will also receive pembrolizumab Day 1 of each cycle beginning with Cycle 2.

For IV cholangiocarcinoma expansion cohort, patients will be treated with CF33-hNIS on Day 3 and Day 17 of each 28 day cycle along with a modified FOLFOX regimen.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patient or legally authorized representative
* Age ≥ 18 years old on the date of consent
* IT/IV cohorts: Any metastatic or advanced solid tumor with documented radiological progression following at least two prior lines of treatment (which may have included prior immune checkpoint inhibitor (ICI) treatment). Expansion cholangiocarcinoma IT and IV cohorts: one prior line of chemotherapy in metastatic/advanced setting. Patients with targetable tumor mutations must have also received 1 line of approved targeted therapy.
* Expansion cholangiocarcinoma IV cohort: prior treatment with leucovorin calcium, fluorouracil, or oxaliplatin is not permitted.
* ECOG performance status 0 - 2
* At least one measurable lesion
* For IT administration, ideally < 5 total lesions no greater than 10cm and <33% of liver volume replaced by tumor.
* Adequate renal function
* Adequate liver function
* Adequate hematologic function
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Prior treatment with a poxvirus based oncolytic virus.
* Continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks prior to first dose of study treatment.
* Prior radiotherapy within 2 weeks of start of study treatment.
* Active autoimmune disease
* Prior allogenic tissue/organ transplant or other medical conditions requiring ongoing treatment with immunosuppressive drugs or any condition resulting in a systemic immunosuppressed state
* Inadequate pulmonary function per Investigator assessment.
* Uncontrolled brain or other central nervous system (CNS) metastases.
* History of documented congestive heart failure (New York Heart Association [NYHA] class III - IV), unstable angina, poorly controlled hypertension, clinically significant valvular heart disease or high-risk uncontrolled arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events of IV and IT CF33-hNIS as a monotherapy or in combination with pembrolizumab | From first dose of study drug through 30 days following the last dose of study treatment.
  Adverse events will be graded according to CTCAE v5.0.
Recommended Phase 2 Dose (RP2D) of CF33-hNIS as a monotherapy or in combination with pembrolizumab | From first dose of study drug through 21-42 days following the first dose of study treatment.
  RP2D determination will be based on evaluation of Dose Limiting Toxicities (DLT) as well as other safety, efficacy and correlative data.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of CF33-hNIS administered as a monotherapy or in combination with pembrolizumab or modified FOLFOX | Up to 2 years from first dose of study drug.
  ORR is defined as the proportion of patients in the efficacy population who achieve a radiographic Investigator-assessed confirmed complete response (CR) or partial response (PR), per RECIST v1.1 or confirmed immune complete response (iCR) or immune partial response (iPR) per iRECIST v1.0.
Progression-free survival (PFS) of CF33-hNIS administered as a monotherapy or in combination with pembrolizumab or modified FOLFOX | Up to 2 years from first dose of study drug.
  PFS, defined as the time from start of treatment to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first.
Overall survival (OS) of CF33-hNIS administered as a monotherapy or in combination with pembrolizumab or modified FOLFOX | Up to 2 years from first dose of study drug.
  defined as the time from the start of treatment until death due to any cause. Median OS and OS rate at 12 months will be reported.
Duration of Response (DOR) of CF33-hNIS administered as a monotherapy or in combination with pembrolizumab or modified FOLFOX | Up to 2 years from first dose of study drug.
  DOR is defined as the time from the date a response of PR/iPR or better was first recorded to the date on which progressive disease was first noted or the date of death due to any cause.
Disease Control Rate (DCR) of CF33-hNIS administered as a monotherapy or in combination with pembrolizumab or modified FOLFOX | Up to 2 years from first dose of study drug.
  DCR is defined as the proportion of patients who achieve an Investigator-assessed confirmed CR/iCR, PR/iPR, or Stable Disease (SD)/immune SD (iSD) per RECIST v1.1 and iRECIST v1.0.
To evaluate viral titers of CF33-hNIS | Up to 2 years from first dose of study drug.
  Viral Plaque Assay (VPA) and polymerase chain reaction (PCR) testing from serum, urine, oral swab, rectal swab, injection site(s) swab and wound dressing swab.
To evaluate infection of tumors with CF33-hNIS | 21 days from first dose of study drug
  hNIS-based imaging via SPECT technetium-99 (99TC).

OTHER OUTCOMES:
To evaluate antiviral immune activation | Up to 2 years from first dose of study drug.
  Up regulation of PD-L1 expression as compared to baseline in tumor tissue and circulating tumor cells (CTC).
  Analysis of lymphocyte subsets and cytokine profile compared to baseline.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology, Springdale, Arkansas
  - City of Hope Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Miami, Miami, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Oncology, Fairfax, Virginia
- Australia (2):
  - Tasman Oncology Research, Southport, Queensland
  - St. Vincent's Hospital, Fitzroy, Victoria

REFERENCES:
- See also: Imugene Limited (ASX: IMU) is a publicly-listed Australian biotechnology company developing cancer immunotherapies. — http://www.imugene.com